CLINICAL TRIAL: NCT03272906
Title: Clinical Feasibility of Transcranial Direct Current Stimulation [tDCS] With Standard Aphasia Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University and A&M College (Other)
Responsible Party: Principal Investigator, E. Susan Duncan, Assistant Professor, Louisiana State University and A&M College
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LEQSF(2017-20)-RD-A-03
Record Dates: First submitted 2017-09-02; First posted 2017-09-06 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Aphasia; Stroke
Keywords: aphasia; stroke; tDCS; language; stimulation; brain; speech therapy
MeSH Terms: conditions — Aphasia; Stroke; Language; Communication Disorders | interventions — Transcranial Direct Current Stimulation; Speech Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- A-tDCS & speech-language therapy (Experimental): Anodal transcranial direct current stimulation (2 mA) plus speech-language therapy for 16 sessions (20-minutes per each 60-minute treatment session) over the course of 8 weeks. The electrical current will be administered over ventral inferior frontal gyrus. The stimulation will be delivered at an intensity of 2mA for a maximum of 20 minutes.
  Interventions: Device: Anodal transcranial direct current stimulation; Behavioral: Speech-language therapy
- Sham-tDCS & speech-language therapy (Sham Comparator): Sham transcranial direct current stimulation (2 mA) plus speech-language therapy for 16 sessions (20-minutes per each 60-minute treatment session) over the course of 8 weeks. Electrodes will be placed as in A-tDCS. Current will be ramped up for the first 30 seconds following which the intensity will drop to 0 mA.
  Interventions: Device: Sham transcranial direct current stimulation; Behavioral: Speech-language therapy

INTERVENTIONS:
Device: Anodal transcranial direct current stimulation — 2 mA of A-tDCS stimulation is induced between two 5 cm x 7 cm saline soaked sponges where one sponge (anode: A-tDCS) is placed on the scalp over the targeted cortical region. Ramping up of the current to 2 mA occurs over 30 seconds to allow participants to habituate to the tingling sensation. A-tDCS stimulation will be active only in the first 20 minutes of the 60-minute treatment session.
  Other Names: (A-tDCS)
  Arms: A-tDCS & speech-language therapy
Device: Sham transcranial direct current stimulation — 2 mA of A-tDCS stimulation is induced between two 5 cm x 7 cm saline soaked sponges where one sponge (anode: A-tDCS) is placed on the scalp over the targeted cortical region. Ramping up of the current to 2 mA occurs over 30 seconds to allow participants to habituate to the tingling sensation. Then, the current will be ramped back down to 0 mA in the sham condition.
  Other Names: Sham
  Arms: Sham-tDCS & speech-language therapy
Behavioral: Speech-language therapy — Therapy tasks will be determined by the clinician on an individualized basis and will not be affected by this research protocol. The only difference between the clinical therapy that is normally provided in the clinic and this research paradigm is the application of tDCS electrodes during therapy. Therapist is blinded to stimulation type.
  Other Names: SLT

SUMMARY:
Study Design: This is a within-subjects crossover design. Subjects will participate in the procedures twice, once under each condition (active vs. sham stimulation). The order of conditions will be counter-balanced across subjects. Stimulation will target ventral inferior frontal gyrus (IFG) and will be paired with standard speech-language therapy. Outcome measures will be acquired at the beginning and end of a semester of standard speech-language therapy.

DETAILED DESCRIPTION:
Baseline Behavioral Assessment: Medical and neurological history will be taken. Western Aphasia Battery-Revised, Communication Activities of Daily Living-2, and Philadelphia Naming Test (short form) will be administered. Narrative will be elicited (Cinderella story). Some of these procedures will be videorecorded for later transcription. Subjects will also complete a pre-tDCS safety screening questionnaire.

tDCS: Participants will undergo placement of 2 tDCS electrodes. For all subjects, the anodal electrode will be placed at the following locations (EEG 10-20 system):

(i) over the left inferior frontal gyrus (crossing point between T3-Fz and F7-Cz)

The cathodal electrode will be placed at the second site:

(ii) over right frontal pole (Fp2)

Two types of stimulation will be given, an active condition and a sham condition. In the sham condition, stimulation is ramped up over the first 30 seconds (as in the active condition), but then discontinued. This gives the physical perception of stimulation without the modulatory effects.

Stimulation will be delivered by a tDCS device with the following parameters for intensity and duration:

* Intensity: 2 mA
* Duration: 20 minutes

tDCS will be provided for the first 20 minutes of each aphasia therapy session provided at the LSU Speech-Language-Hearing Clinic. The therapy sessions last for one hour and are provided twice weekly for 8 weeks over the course of an academic semester (fall and spring).

Post-Therapy/Stimulation Assessment: Western Aphasia Battery-Revised, Communication Activities of Daily Living-2, and Philadelphia Naming Test (short form) will be administered as before therapy. Cinderella narrative will again be elicited. Some of these procedures will again be videorecorded for later transcription. A tDCS sensations survey will also be completed at the final assessment to determine the effectiveness of blinding.

ELIGIBILITY:
Inclusion Criteria:

* Single, unilateral stroke resulting in aphasia
* Competency to provide written informed consent
* Ability to participate in standard aphasia therapy

Exclusion Criteria:

* Serious psychological condition
* Serious neurological condition, other than stroke
* Serious medical condition
* Pregnancy
* History of seizures
* Presence of electronic or metal implants (e.g., pacemaker, vagal nerve stimulator, etc.).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Production of Correct Information Units (CIUs) in Cinderella narrative | Following 8 weeks of speech-language therapy
  Change in CIU production over treatment interval. Words are counted as CIUs if they are novel, intelligible, and appropriate in context

SECONDARY OUTCOMES:
Western Aphasia Battery-Revised (WAB-R) | Following 8 weeks of speech-language therapy
  Change in performance on Part 1 of WAB-R (Aphasia Quotient)
Communication Activities of Daily Living-2 (CADL-2) | Following 8 weeks of speech-language therapy
  Change in performance on CADL-2
Philadelphia Naming Test - Short Form (PNT) | Following 8 weeks of speech-language therapy
  Change in performance on PNT

CONTACTS AND LOCATIONS:
Overall Officials: E. Susan Duncan, PhD, CCC-SLP, Principal Investigator — Lousiana State University
Locations (1):
- Louisiana State University, Baton Rouge, Louisiana, United States